CLINICAL TRIAL: NCT06365671
Title: A Single-Arm Clinical Study of CD19 CAR-T Following ASCT for Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma (R/R B-NHL) With High-Risk Prognostic Factors
Brief Title: CAR-T Following ASCT for Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma (R/R B-NHL) With High-Risk Prognostic Factors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASCT-CART
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T following ASCT (Experimental): Participants will receive high-dose chemotherapy followed by stem-cell infusion, and a fixed dose of CAR-T cells will be infused.
  Interventions: Other: autologous stem-cell transplantation; Drug: Relmacabtagene autoleucel (relma-cel)

INTERVENTIONS:
Other: autologous stem-cell transplantation — high-dose chemotherapy and autologous stem-cell transplantation (HDT/ASCT)
Drug: Relmacabtagene autoleucel (relma-cel) — relma-cel (CD19 CAR-T cell)infusion on day 3(±1d) after ASCT with a fixed dose of 100X10^6.

SUMMARY:
Clinical trial for the safety and efficacy of CD19 CAR-T following autologous hematopoietic stem cell transplantation (ASCT) for Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma (R/R B-NHL) with High-Risk Prognostic Factors

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label, prospective clinical trial to evaluate the efficacy and safety of CD19 CAR-T infusion following high-dose chemotherapy and autologous stem-cell transplantation (HDT/ASCT) in relapsed or refractory B-cell Non-Hodgkin's Lymphoma patients with high-risk prognostic factors (extranodal involvement/bulky mass ≥5 cm in diameter/TP53 alterations). CD19 CAR-T will be infused on day +3 (±1d) with a fixed dose of 100X10^6. The study will assess the safety and efficacy of this combinational therapy, including the investigators assessed the best complete response rate (BCR) in 3 months (primary endpoint), objective response rates, survivals, incidence and severity of cytokine release syndrome (CRS), immune effector cell-associated neurotoxicity syndrome (ICANS), hematological, and other non-hematological toxicities of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed B-cell non-Hodgkin's lymphoma including the following types

   * diffuse large B-cell lymphoma
   * high-grade B-cell lymphoma with or without MYC and BLC2 and/or BCL6 rearrangement
   * transformed lymphoma
   * primary mediastinal large B-cell lymphoma
   * follicular lymphoma (FL)
2. Relapsed or refractory diseases fulfilling one of the following criteria (individuals must have received anti-CD20 monoclonal antibody and anthracycline-containing chemotherapy regimen)

   * Primary refractory disease, defined as disease progression after first-line immunochemotherapy or disease progression within 6 weeks of the end of the last chemotherapy
   * Stable disease (SD) as best response after at least 4 cycles of first-line therapy
   * Partial response (PR) as best response after at least 6 cycles of first-line therapy (biopsy-proven residual disease is needed for individuals with Deauville score of 4)
   * PR as best response after at least 2 cycles of second-line therapy
   * Disease relapse ≤12 months after the completion of first-line immunochemotherapy
   * Relapsed or refractory disease after ≥2 lines of chemotherapy
3. Presence of at least one of the following high-risk prognostic factors: (1) extranodal involvement; (2) maximum diameter of the bulky mass ≥5 cm; (3) TP53 gene alterations
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
5. Eligible for HDCT/ASCT based on the investigator's assessment and are scheduled to undergo an ASCT sequential CAR-T treatment regimen
6. Adequate renal and hepatic function defined as:

   * Serum alanine aminotransferase (ALT/AST) ≤ 3 upper limit of normal (ULN)
   * Total bilirubin ≤1.5 mg/dL(<3 times ULN in patients with Gilbert's syndrome, cholestasis due to hepatoportal compression adenopathy, biliary obstruction in patients with liver involvement or lymphoma)
   * Serum creatinine ≤1.5 ULN, or creatinine clearance (as estimated by Cockcroft Gault) ≥ 30 mL/min
7. Cardiac ejection fraction ≥ 40%
8. Baseline oxygen saturation > 95% on room air
9. Life expectancy ≥3 months

Exclusion Criteria:

1. History of autologous or allogeneic stem cell transplantation
2. Active HBV or HCV infection, defined as HBV-DNA or HCV-DNA levels above the normal upper limit, with or without abnormal liver function. Individuals with positive HBsAg or HBcAb should receive antiviral prophylaxis for at least 12 months after CAR-T cells infusion.
3. Presence of uncontrolled infection, cardio-cerebrovascular disease，coagulopathy, or connective tissue disease.
4. History of HIV infection
5. Prior chimeric antigen receptor cellular immunotherapy targeting CD19
6. Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Best Complete Response (CR) Rate in 3 months | 3months post CAR-T infusion
  Best Complete Response rate in 3 months is defined as the incidence of subjects achieving complete remission (CR) within 3 months after CAR-T infusion according to the Lugano Classification (Cheson et al, 2014), as determined by study investigators.

SECONDARY OUTCOMES:
Objective remission rate (ORR) in 3months | 3months post CAR-T infusion
  ORR in 3 moths is defined as the incidence of either a CR or a partial response (PR) within 3 months after CAR-T infusion per the Lugano Classification as determined by study investigators.
Duration of Response (DOR) | 2 years post CAR-T infusion
  DOR is defined only for participants who experience an objective response after CAR-T infusion and is the time from the first objective response to disease progression or death from any cause
Progression-Free Survival (PFS) | 2 years post CAR-T infusion
  PFS is defined as the time from the CAR-T infusion date to the date of disease progression or death from any cause.
Overall Survival (OS) | 2 years post CAR-T infusion
  OS is defined as the time from CAR-T infusion to the date of death from any cause.
Adverse Events rate as assessed by CTCAE version 5.0 | 2 years post CAR-T infusion
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China